CLINICAL TRIAL: NCT04482881
Title: Isosorbide Mononitrate and Misoprostol in Induction of Labour
Brief Title: Isosorbide Mononitrate in Induction of Labour
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: labour induction
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Labor Fast
MeSH Terms: interventions — isosorbide-5-mononitrate; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- women receiving isosorbide mononitrates lower dose (Active Comparator): women who will receive isosorbide mononitrates lower dose
  Interventions: Drug: Isosorbide Mononitrate 40 MG
- women receiving isosorbide mononitrates higher dose (Active Comparator): women who will receive isosorbide mononitrates higher dose
  Interventions: Drug: Isosorbide Mononitrate 60 MG
- Women receiving misoprostol (Active Comparator): Women who will receive misoprostol
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Isosorbide Mononitrate 40 MG — giving women isosorbide mononitrate 40 MG
  Arms: women receiving isosorbide mononitrates lower dose
Drug: Isosorbide Mononitrate 60 MG — giving women isosorbide mononitrate 60MG
  Arms: women receiving isosorbide mononitrates higher dose
Drug: Misoprostol — Giving women misoprostol
  Arms: Women receiving misoprostol

SUMMARY:
Induction of labor is defined as the process of artificially initiating uterine contractions, prior to their spontaneous onset, with progressive effacement and dilatation of the cervix and ultimately, the delivery of the baby.

DETAILED DESCRIPTION:
There are many indications for induction of labor in the obstetric practice, of which prolonged gestational age stands as the most common cause.

ELIGIBILITY:
Inclusion Criteria:

* Single vertex presentation. 2. Gestational age > 37weeks calculated from last menstrual period or U/S scanning.

Exclusion Criteria:

1. Patients with rupture of membranes.
2. Previous uterine scar.
3. Fetal malpresentation.
4. Multiple pregnancies.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 130 (Estimated)
Dates: Start 2020-07-21 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
the number of women who will be reach active phase within 24 hours | 24 hours
  how many women will reach active phase within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah, Giza, Egypt